CLINICAL TRIAL: NCT01656824
Title: Study of Human Primary Cancer Tissue Implanted in Mice Lacking Bv8/PH-2 in Their Bone Marrow-derived Cells
Brief Title: Tissue Study of Bv8/PK-2 Inhibition in Human Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Other Study IDs: Bv8/PK-2CTIL
Record Dates: First submitted 2012-08-01; First posted 2012-08-03 (Estimated); Last update posted 2013-11-21 (Estimated); Status verified 2013-11

CONDITIONS: Cancer
Keywords: Bv8/PK-2; MDSC Myeloid Derived Suppressor Cells; BMDC Bone Marrow Derived Cells; Angiogenesis; Pancreatic Cancer
MeSH Terms: conditions — Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Biospecimen Retention: Samples With DNA — cancer tissues
Oversight: Data Monitoring Committee: No

SUMMARY:
Study hypothesis is that inhibition of Bv8 production in bone marrow cells of a mice wil reduce the rate of growth of a primary human tumor implanted in the mice. we will take mice and transform their bone marrow cells into non-Bv8 producing cells. than we will implant primary human tumor tissue (taken from surgical specimens after informed consent)in those mice and follow-up on the mice.

DETAILED DESCRIPTION:
1-10 grams of human cancer tissue will be taken from surgical specimen without interference to the pathological data gathering process. those tissues will be implanted in nude mice that will either be treated with anti-Bv8 antibodies or will be transplanted with bone marrow in which Bv8 expression is silenced.

ELIGIBILITY:
Inclusion Criteria:

* ages 18-85 years
* Pathologically-confirmed diagnosis of pancreatic ductal adenocarcinoma undergoing surgical pancreaticoduodenectomy

Exclusion Criteria:

* refuse to take part
* preoperative chemotherapy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with pancreatic cancer and are candidates for whipple's procedure
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2012-08; Primary Completion 2014-09 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Tumor growth in xenograft model | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Erez Hasnis, MD;PhD, Principal Investigator — Rambam Health Care Campus; Erez Hasnis, MD; PhD., Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Medical Center, Haifa, Israel